CLINICAL TRIAL: NCT01533727
Title: A Phase 2,Open-label Study of Autologous Cytokine-Induced Killer Cell Transfusion Plus Chemotherapy as Adjuvant Therapy for Stage IB-IIIA Non-Small Cell Lung Cancer
Brief Title: CIK Cell Transfusion Plus Chemotherapy as Adjuvant Therapy for Stage IB-IIIA Non-Small Cell Lung Cancer (NSCLC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Few patients would like to participate ,since CIK cell transfusion was a new treatment and its efficacy was doubted.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010014
Record Dates: First submitted 2012-02-12; First posted 2012-02-15 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2012-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Cytokine-Induced Killer Cell; NSCLC; adjuvant therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Autologous CIK Transfusion plus Chemotherapy
  Interventions: Drug: Autologous CIK Transfusion plus Chemotherapy
- Group B (Active Comparator): chemotherapy alone
  Interventions: Drug: chemotherapy alone

INTERVENTIONS:
Drug: Autologous CIK Transfusion plus Chemotherapy — vinorelbine 25-30mg/m2 d1, d8 q3w; DDP 75mg/m2 d1 q3w; pemetrexed 500mg/m2 d1 q3w; carboplatin AUC 5/6 q3w; CIK infusion D14 q3w
  Arms: Group A
Drug: chemotherapy alone — vinorelbine 25-30mg/m2 d1, d8 q3w; DDP 75mg/m2 d1 q3w; pemetrexed 500mg/m2 d1 q3w; carboplatin AUC 5/6 q3w;
  Arms: Group B

SUMMARY:
Non - small cell lung cancer ( NSCLC ) accounts for more than 80% of lung cancer. The main treatment for early stage patients is surgical resection, but about 30% -70% patients will relapse. Postoperative chemotherapy is the major systemic treatment for surgical resection NSCLC patients. However, data show only 5-10% improvement in overall survival with systemic adjuvant chemotherapy. It is necessary to further improve the survival time of patients with lung cancer. Biological treatment is becoming a new treatment modality for Cancer following with surgery, radiotherapy and chemotherapy, and has been confirmed as an effective adjuvant treatment in comprehensive cancer treatment. Cytokine induced killer cells ( CIK) characterized as fast amplification, strong anti-cancer activity and broad anti-tumor spectrum is most widely used and thought to be the first choice for the new generation of anti-tumor adoptive immunotherapy. This Phase II study is investigating the efficacy of Autologous Cytokine-Induced Killer Cell Transfusion plus Chemotherapy as adjuvant therapy for stage IB-IIIA NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IB-IIIA post-surgery NSCLC patients with histologically confirmed.
2. with an Eastern CooperativeOncology Group performance status of 0 or 1,
3. at least 18 years of age
4. adequate bone marrow reserve and organ function including calculated creatinine clearance 45 mL/min based on the standard Cockcroft and Gault formula
5. patients had fully recovered from its acute effects.

Exclusion Criteria:

1. HIV positive
2. autoimmune disease
3. immune deficiency disorder
4. organ transplantation
5. received high dose glucocorticoid or other immune depressant within 4 weeks
6. active clinically serious infections (> grade 2 NCI-CTC version 3.0)
7. life threatening medical condition

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2017-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
the relapse rate | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China